CLINICAL TRIAL: NCT00030446
Title: A Phase II Study Of OSI-774 (NSC 718781) Given In Combination With Carboplatin In Patients With Recurrent Epithelial Ovarian Cancer
Brief Title: Erlotinib and Carboplatin in Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I149; CAN-NCIC-149 (Other: PDQ); CDR0000069166 (Other: PDQ)
Record Dates: First submitted 2002-02-14; First posted 2003-06-27 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Drug: carboplatin
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib with carboplatin may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining erlotinib and carboplatin in treating patients who have recurrent ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer treated with erlotinib and carboplatin.
* Determine the duration of stable disease, time to progression, and response duration in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Correlate the level of epidermal growth factor receptor tumor expression with objective tumor response in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to response to prior platinum-containing therapy (platinum-sensitive, defined as 6 months or more since prior therapy with platinum agent [closed to accrual as of 2/13/2004], vs platinum-resistant, defined as less than 6 months since prior therapy with platinum agent).

Patients receive carboplatin IV over 30 minutes on day 1 and oral erlotinib once daily on days 1-21. Treatment repeats every 21 days for up to 6 courses. After the completion of 6 courses of therapy, patients with responsive or stable disease may continue to receive erlotinib and carboplatin in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 23-60 patients (8-30 for platinum-sensitive stratum [closed to accrual as of 2/13/2004] and 15-30 for platinum-resistant stratum) will be accrued for this study within 15-23 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent ovarian epithelial, fallopian tube, or primary peritoneal cancer for which no standard curative therapy exists
* At least 1 measurable lesion

  * At least 20 mm by x-ray, non-spiral CT scan, or physical exam OR at least 10 mm by spiral CT scan
  * Ascites and bone metastases not considered measurable disease
* No abdominal adenocarcinoma of unknown origin or borderline ovarian tumor
* No elevated CA 125 as only evidence of disease
* At least 1 but no more than 2 prior chemotherapy regimens required

  * First regimen must have contained cisplatin or carboplatin
  * Switching platinum compounds due to disease progression or failure to respond is considered 2 regimens
  * Same regimen as first- and second-line therapy is considered 2 regimens
* Responded to prior platinum-based first-line chemotherapy

  * No platinum-refractory disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than ULN

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina
* No cardiac arrhythmia

Gastrointestinal:

* See Surgery
* No GI tract disease resulting in an inability to take oral medication or requiring IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* No active peptic ulcer disease

Ophthalmic:

* No ocular inflammation or infection
* No significant ophthalmologic abnormalities, including:

  * History of dry eye syndrome, Sjögren's syndrome, or keratoconjunctivitis sicca
  * Severe exposure keratopathy
  * Disorders that might increase the risk for epithelium-related complications (e.g., bullous keratopathy, aniridia, severe chemical burns, or neutrophilic keratitis)
  * Congenital abnormality (e.g., Fuch's dystrophy)
  * Abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
  * Abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reaction to compounds of similar chemical or biological composition to erlotinib
* No other serious illness, medical condition, or significant neurologic or psychiatric disorder that would preclude study therapy
* No active uncontrolled infection
* No grade 3 or greater drug-related neurotoxicity
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since prior radiotherapy (except low-dose palliative radiotherapy) and recovered

Surgery:

* At least 3 weeks since prior major surgery (wound healing must have occurred)
* No prior surgical procedures affecting gastrointestinal (GI) absorption
* No concurrent ophthalmic surgery

Other:

* No prior therapy targeting epidermal growth factor receptor
* No other concurrent anticancer therapy
* No other concurrent investigational agents
* Concurrent oral anticoagulants (e.g., warfarin) allowed provided INR is monitored

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-01-10 (Actual); Primary Completion 2005-02-11 (Actual); Study Completion 2009-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hal W. Hirte, MD, FRCP(C), Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (8):
- Canada (8):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre- Dame du CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hirte H, Oza A, Hoskins P, et al.: Phase II study of OSI-774 given in combination with carboplatin in patients (pts) with recurrent epithelial ovarian cancer (EOC): NCIC CTG IND.149. [Abstract] European Journal of Cancer Supplements 1 (5): A-159, S51, 2003.